CLINICAL TRIAL: NCT03050749
Title: A Prospective, Open-label, Non-comparative, Multicentre, Post-market Clinical Follow-up Study of the Princess® VOLUME Performance and Safety for Correction of Facial Lipoatrophy, Morphological Asymmetry of the Face, or Debilitating Scars
Brief Title: Safety and Performance of Princess® VOLUME for the Treatment of Facial Lipoatrophy, Asymmetry or Scars
Acronym: FLASH2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CPH-401-201260
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Facial Lipoatrophy; Morphological Asymmetry of the Face; Debilitating Scars

STUDY DESIGN:
Intervention Model Description: Princess® VOLUME
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Princess® VOLUME (Other)
  Interventions: Device: Princess® VOLUME

INTERVENTIONS:
Device: Princess® VOLUME — Princess® VOLUME injections up to 10 ml applied to the eligible subjects at the baseline visit, and the touch-up visit, if applicable.

SUMMARY:
In this study, eligible patients with the medical indications (facial lipoatrophy, morphological asymmetry of the face, or debilitating scars) will be treated with Princess® VOLUME, and then will return for follow-up assessments 2, 4, 24, and 36 weeks after the treatment. A touch-up treatment may be done 2 weeks after the treatment if deemed appropriate by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* Presence of a defect, which in the opinion of the Investigator can be corrected by a dermal filler, and is caused by: ° Facial lipoatrophy of moderate severity, or

  * Morphological asymmetry of the face, or
  * One or more debilitating scars on the face
* Willingness to abstain from any cosmetic or surgical procedures in the treatment area for the duration of the clinical investigation
* Willingness to take part in the clinical investigation as evidenced by a personally signed informed consent.

Exclusion Criteria:

* Pregnancy, breastfeeding, or unwillingness to use contraception throughout the clinical investigation (for women of child-bearing potential only)
* History of allergic reaction or hypersensitivity to hyaluronic acid
* History or presence of any autoimmune or connective tissue disease, or current treatment with immune therapy
* Presence of silicone implant or other non-absorbable tissue filler in the area targeted for intervention, or pre-treatment with any hyaluronic acid filler within the last six months
* Presence of infectious, inflammatory, or proliferative lesions in the area targeted for intervention
* Treatment with anticoagulant or antiplatelet drugs
* Any disease or condition which, in the Investigator's opinion, represents a safety risk for participation in the study
* Current participation in another clinical trial, or previous treatment with any investigational drug/device within 30 days prior to enrolment
* Institutionalized persons with legally limited civil rights

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-11-20 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
6-point scale for clinical response | 4 week
  The proportion of patients with successful treatment outcome at the Week 4 visit based on the Investigator's opinion, where success is defined as excellent, good, or moderate correction of the defect

CONTACTS AND LOCATIONS:
Overall Officials: Daisy Kopera, Prof., Principal Investigator — Medical University Graz, Austria
Locations (3):
- Austria (3):
  - Medical University Graz, Graz
  - MÄZ WIEN Medizinisch Ästhetisches Zentrum Wien, Vienna
  - Ordination Dr. Benjamin Gehl, Vienna

IPD SHARING:
Plan to Share IPD: No